CLINICAL TRIAL: NCT03106623
Title: Phase 2a Exploratory, Randomized, Double-blind, Parallel-group Study of ONO-8577 Compared to Combination of Solifenacin Succinate/ Mirabegron for Overactive Bladder
Brief Title: Study of ONO-8577 in Patients With Overactive Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ONO-8577-02
Record Dates: First submitted 2017-03-15; First posted 2017-04-10 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate; mirabegron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ONO-8577 Arm (Experimental): Oral administration of ONO-8577 once a daily for 4 weeks
  Interventions: Drug: ONO-8577
- Active Comparator Arm (Active Comparator): Oral administration of solifenacin succinate and mirabegron once a daily for 4 weeks
  Interventions: Drug: solifenacin succinate + mirabegron
- Placebo Arm (Placebo Comparator): Oral administration of Placebo once a daily for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ONO-8577 — Oral administration of ONO-8577 once a daily for 4 weeks
  Arms: ONO-8577 Arm
Drug: solifenacin succinate + mirabegron — Oral administration of solifenacin succinate and mirabegron once a daily for 4 weeks
  Arms: Active Comparator Arm
Drug: Placebo — Oral administration of Placebo once a daily for 4 weeks
  Arms: Placebo Arm

SUMMARY:
The objective of the study is to evaluate the efficacy and safety of ONO-8577 compared to combination of solifenacin succinate and mirabegron or placebo for overactive bladder

ELIGIBILITY:
Inclusion Criteria:

* Patient with symptoms of overactive bladder for ≥6 months

Exclusion Criteria:

* Patient with genuine stress incontinence, or with stress-predominant mixed urinary incontinence
* Patient who has never experienced urge urinary incontinence during disease duration of overactive bladder

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2017-09-26 (Actual)

PRIMARY OUTCOMES:
Efficacy (Change From Baseline to Week 4 in Mean Number of Micturitions Per 24 Hours) | Baseline and Week 4

SECONDARY OUTCOMES:
Safety (adverse event, vital signs, 12-lead electrocardiography, residual urine volume, clinical laboratory test) | Up to Week 4
Pharmacokinetics (plasma concentration at one point on each visit) | Week 2 and 4
Efficacy (Change From Baseline to Week 2 in Mean Number of Micturitions Per 24 Hours) | Baseline and Week 2
Efficacy (Change and Change Rate From Baseline to Week 2 and 4 in Mean Number of Micturitions Per 24 Hours) | Baseline, Week 2 and 4
Efficacy (Change and Change Rate From Baseline to Week 2 and 4 in Mean Number of Incontinence Episodes Per 24 Hours) | Baseline, Week 2 and 4
Efficacy (Change and Change Rate From Baseline to Week 2 and 4 in Mean Number of Urgency Incontinence Episodes Per 24 Hours) | Baseline, Week 2 and 4
Efficacy (Change and Change Rate From Baseline to Week 2 and 4 in Mean Number of Urgency Episodes Per 24 Hours) | Baseline, Week 2 and 4
Efficacy (Change and Change Rate From Baseline to Week 2 and 4 in Mean Number of Nocturia Episodes Per 24 Hours) | Baseline, Week 2 and 4
Efficacy (Percentage of Participants With ˂8 times of Micturitions Per 24 Hours at Week 2 and 4) | Week 2 and 4
Efficacy (Percentage of Participants With Zero Incontinence Episodes at Week 2 and 4 | Week 2 and 4
Efficacy (Change and Change Rate From Baseline to Week 2 and 4 in Mean Volume Voided Per Micturition) | Baseline, Week 2 and 4
Efficacy (Change From Baseline to Week 2 and 4 in Overactive Bladder Symptom Score (OABSS) ) | Baseline, Week 2 and 4
Efficacy (Change From Baseline to Week 4 in Health-related Quality of Life) | Baseline and Week 4
Efficacy (Patient Global Impression at Week 4) | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Hitoshi Kajitani, Study Director — Ono Pharmaceutical Co. Ltd
Locations (30):
- Japan (30):
  - Gunma Clinical Site 02, Maebashi, Gunma
  - Gunma Clinical Site 01, Takasaki, Gunma
  - Hyogo Clinical Site 02, Akashi, Hyōgo
  - Hyogo Clinical Site 01, Kobe, Hyōgo
  - Hyogo Clinical Site 03, Kobe, Hyōgo
  - Hyogo Clinical Site 04, Takarazuka, Hyōgo
  - Kanagawa Clinical Site 01, Isehara, Kanagawa
  - Kanagawa Clinical Site 02, Kamakura, Kanagawa
  - Kanagawa Clinical Site 03, Sagamihara, Kanagawa
  - Kanagawa Clinical Site 04, Yokohama, Kanagawa
  - Osaka Clinical Site 03, Higashiosaka, Osaka
  - Osaka Clinical Site 04, Ibaraki, Osaka
  - Osaka Clinical Site 02, Osaka, Osaka
  - Osaka Clinical Site 05, Suita, Osaka
  - Osaka Clinical Site 06, Toyonaka, Osaka
  - Osaka Clinical Site 07, Toyonaka, Osaka
  - Saitama Clinical Site 01, Kumagaya, Saitama
  - Osaka Clinical Site 01, Osaka, Takatsuki-shi
  - Tokyo Clinical Site 10, Bunkyo-ku, Tokyo
  - Tokyo Clinical Site 01, Edogawa-ku, Tokyo
  - Tokyo Clinical Site 06, Itabashi-ku, Tokyo
  - Tokyo Clinical Site 09, Nakano-ku, Tokyo
  - Tokyo Clinical Site 07, Nerima-ku, Tokyo
  - Tokyo Clinical Site 03, Ōta-ku, Tokyo
  - Tokyo Clinical Site 08, Setagaya-ku, Tokyo
  - Tokyo Clinical Site 11, Setagaya-ku, Tokyo
  - Tokyo Clinical Site 04, Shinagawa-ku, Tokyo
  - Tokyo Clinical Site 05, Shinagawa-ku, Tokyo
  - Tokyo Clinical Site 02, Suginami-ku, Tokyo
  - Kyoto Clinical Site 01, Kyoto

IPD SHARING:
Plan to Share IPD: No